CLINICAL TRIAL: NCT03838042
Title: INFORM2 Exploratory Multinational Phase I/II Combination Study of Nivolumab and Entinostat in Children and Adolescents With Refractory High-risk Malignancies (INFORM2-NivEnt)
Brief Title: INFORM2 Study Uses Nivolumab and Entinostat in Children and Adolescents With High-risk Refractory Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Olaf Witt, MD, Prof. Dr. Olaf Witt, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Final4, 18-10-2023; 2018-000127-14 (EudraCT Number); NCT-2017-0516 (Other: Sponsor's No)
Record Dates: First submitted 2019-02-04; First posted 2019-02-12 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: CNS Tumor; Solid Tumor
Keywords: high-risk solid tumors; high-risk CNS tumors
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Nivolumab; entinostat

STUDY DESIGN:
Intervention Model Description: Phase I:
  To determine the recommended phase II dose (RP2D) of the combination treatment with nivolumab and entinostat administered to adolescents 12-21 years with progressive, relapsed, refractory high-risk solid tumors and CNS tumors To determine the recommended phase II dose (RP2D) of the combination treatment with nivolumab and entinostat administered to children 6-11 years with progressive, relapsed, refractory high-risk solid tumors and CNS Tumors
  Phase II:
  To evaluate activity and safety of the combination treatment with nivolumab and entinostat in children and adolescents aged 2-21 years with refractory/relapsed/progressive high-risk solid tumors and CNS tumors with:
  Group A: a high mutational load (> 100 somatic SNVs/exome), Group C: Focal MYC(N) amplification or ATRT-MYC subgroup, Group E: high TILs or TLS positive (> 600 cells/mm² or presence of TLS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nivolumab and Entinostat (Experimental): Combination Study of Nivolumab and Entinostat
  Interventions: Drug: Nivolumab and Entinostat

INTERVENTIONS:
Drug: Nivolumab and Entinostat — Patients entering phase I will receive one week entinostat without nivolumab (priming phase) before receiving the combination treatment of nivolumab and entinostat.
  Other Names: Opdivo

SUMMARY:
The aim of this trial is to determine preliminary activity of the combination treatment with nivolumab and entinostat in children and adolescents with high risk refractory/relapsed/progressive tumors harboring a high mutational load, focal MYC(N) amplification or ATRT-MYC subgroup as well as tumors with high tumor infiltrating lymphocytes (TILs) or a tertiary lymphoid structure (TLS).

DETAILED DESCRIPTION:
Compared to adult cancers, most pediatric cancers carry a relatively low mutational burden. HDAC inhibition (HDACi) modifies T-cell regulation and can augment response to checkpoint inhibition by reducing the number of myeloid-derived suppressor cells and creating an immunogenic tumor microenvironment including induction of MHCI and neo-antigens. In vitro and in vivo models showed enhanced anti-tumor activity of the combination of checkpoint inhibition and HDACi compared to either agent alone. This provides a strong rationale to combine these drug classes. Checkpoint inhibition results in activation of tumor-associated T cells. It is now becoming increasingly evident that patients with tumors with a high number of tumor infiltrating T cells at baseline show an increased response rate. Additionally, recent clinical data on immune checkpoint inhibition (ICI) for melanoma patients detected tertiary lymphoid structures (TLS) as indicators of an activated adaptive immune response. Their presence has been linked to objective treatment responses in patients with different cancer entities receiving ICI.

Furthermore, MYC- or NMYC-driven (referred to as MYC(N)) malignancies like very high-risk medulloblastomas or very high-risk neuroblastomas still have a dismal outcome. MYC is not only reported to upregulate PD-L1 and thereby a possible biomarker for checkpoint inhibition but also very compelling recent preclinical data strongly suggests that HDAC inhibitors are active against MYC amplified medulloblastoma in vitro and in vivo. In NMYC amplified neuroblastoma cell lines similar observations were made in vitro. In addition, it has been shown recently that the molecular MYC subgroup of atypical teratoid rhabdoid tumors (ATRT) exhibit a strong T-cell infiltrate in contrast to the SHH-ATRT subtype and are considered immunological "hot" tumors. Taken together, our results suggest that MYC(N)-driven tumors depend on HDAC and we hypothesize that MYC(N) status can serve as a biomarker for response prediction to a combinatorial treatment of checkpoint inhibition and HDAC inhibition.

Pediatric patients aged 2-21 years with refractory/relapsed/progressive high-risk malignancies with a high mutational load (group A), with MYC(N) amplification or from the ATRT-MYC subgroup (group C) as well as patients with high TILs and/or TLS positive (group E) are eligible for this trial. Phase I determines the recommended phase 2 dose (RP2D) for the combination of the HDACi entinostat and the checkpoint inhibitor nivolumab for the age groups 6-11 and 12-21 years, respectively. Phase II investigates activity in 3 groups A, C, E for patients in the two age cohorts 2-11 and 12-21 years. The duration of treatment is 12 cycles (1 cycle = 28 days), preceded by 1 priming week.

In addition, a comprehensive accompanying research program investigates PD biomarkers for immune checkpoint and HDAC inhibition.

Clinical trials investigating the combination of nivolumab and entinostat in children have not been reported so far.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with refractory/relapsed/progressive high-risk

  * CNS tumors: medulloblastoma, ependymoma, ATRT, ETMR, pediatric high grade glioma (including DIPG) or other pediatric embryonal CNS tumors OR
  * solid tumors: neuroblastoma, nephroblastoma, rhabdoid tumor, embryonal or alveolar rhabdomyosarcoma, other embryonal small round blue cell tumors including pediatric type (bone) sarcoma or other pediatric type solid tumors OR
  * Children and adolescents with newly diagnosed high grade glioma (HGG) in the context of a constitutional mismatch repair deficiency syndrome after maximum safe surgical resection with no established standard of care treatment option with curative intention available. In addition in France: ineligible to radiotherapy
* No standard of care treatment available
* Age at registration ≥ 2 to ≤ 21 years
* Molecular analysis for biomarker identification (SNV load, MYC/N amplification, high TILs or TLS positive) in laboratories complying with DIN EN ISO/IEC 17025 or similar via INFORM molecular diagnostic platform or equivalently valid molecular pipeline
* Biomarker determined using whole exome sequencing (SNV load), whole genome- or whole exome sequencing (MYC/N amplification), IHC (high TILs or TLS positive)
* In case molecular analysis was not performed via INFORM Registry molecular pipeline: transfer of molecular data (whole exome sequencing)
* Time between biopsy/puncture/resection of the current refractory/relapsed/progressive tumor and registration ≤ 24 weeks. In patients receiving therapy not impacting biomarker stratification, time between biopsy/puncture/resection of the current refractory/relapsed/progressive tumor and registration of ≤ 36 weeks is allowed
* Disease that is measurable as defined by RANO criteria or RECIST v1.1 (as appropriate).
* Life expectancy > 3 months, sufficient general condition score (Lansky ≥ 70 or Karnofsky ≥ 70). Transient states like infections requiring antibiotic treatments can be accepted, and also stable disabilities resulting from disease/surgery (hemiparesis, amputations etc.) can be accepted and will not be considered for Lansky/Karnofsky assessments.
* Laboratory requirements:

  * Hematology:

    * absolute granulocytes ≥ 1.0 × 109/l (unsupported)
    * platelets ≥ 100 × 109/l & stable
    * hemoglobin ≥ 8 g/dl or ≥ 4.96 mmol/L
  * Biochemistry:

    * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
    * AST(SGOT) ≤ 3.0 x ULN
    * ALT(SGPT) ≤ 3.0 x ULN
    * serum creatinine ≤ 1.5 x ULN for age
* ECG: normal QTc interval according to Bazett formula < 440ms
* Patient is able to swallow oral study medication
* Ability of patient and/or legal representative(s) to understand the character and individual consequences of clinical trial
* Females of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to initiation of treatment. Sexually active women of childbearing potential must agree to use acceptable and appropriate contraception during the study and for at least 6 months after the last study treatment administration. Sexually active male patients must agree to use a condom during the study and for at least 3 months after the last study treatment administration.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient screening and registration, written informed consent, also concerning data and blood transfer, must be given according to ICH/GCP, and national/local regulations.
* No prior therapy with the combination of immune checkpoint inhibitors and HDACi
* Phase I: molecular analysis performed and biomarker status known (mutational load, high TILs or TLS positive AND MYC(N) amplification status).
* Phase II: molecular analysis performed, biomarker status known (mutational load, high TILs or TLS positive AND MYC(N) amplification status) and stratification according to the following criteria:

  * Group A: high mutational load (defined as > 100 somatic SNVs/exome) based on whole exome sequencing OR
  * Group C: Focal MYC(N) amplification based on whole genome sequencing or whole exome sequencing ot ATRT-MYC subgroup OR
  * Group E: high TILs or TLS positive (defined as cells per mm² > 600 or presence of tertiary lymphoid structure) based on IHC analysis.

Exclusion Criteria:

* Patients with CNS tumors or metastases who are neurologically unstable despite adequate treatment (e.g. convulsions).
* Patients with low-grade gliomas or tumors of unknown malignant potential are not eligible
* Evidence of > Grade 1 recent CNS hemorrhage on the baseline MRI scan.
* Participants with bulky CNS tumor on imaging are ineligible; bulky tumor is defined as:

  * Tumor with any evidence of uncal herniation or severe midline shift
  * Tumor with diameter of > 6 cm in one dimension on contrast-enhanced MRI
  * Tumor that in the opinion of the investigator, shows significant mass effect
* Previous allogeneic bone marrow, stem cell or organ transplantation
* Diagnosis of immunodeficiency
* Diagnosis of prior or active autoimmune disease
* Evidence of interstitial lung disease
* Any contraindication to oral agents or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the investigator, would preclude adequate absorption.
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies). Known active hepatitis B (e.g., hepatitis B surface antigen-reactive) or hepatitis C (e.g., hepatitis C virus ribonucleic acid [qualitative]). Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible. HBV DNA test must be performed in these patients prior to study treatment. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Clinically significant, uncontrolled heart disease
* Major surgery within 21 days of the first dose. Gastrostomy, ventriculo-peritoneal shunt, endoscopic ventriculostomy, tumor biopsy and insertion of central venous access devices are not considered major surgery, but for these procedures, a 48 hour interval must be maintained before the first dose of the investigational drug is administered.
* Any anticancer therapy (e.g., chemotherapy, HDACi (including valproic acid), DNA methyltransferase inhibitors, other immunotherapy, targeted therapy, biological response modifiers, endocrine anticancer therapy or radiotherapy) within 2 weeks or at least 5 half- lives (whichever is longer) of study drug administration.
* Radiologically confirmed radiotherapy induced pseudoprogression in CNS tumors
* Traditional herbal medicines; these therapies are not fully studied and their use may result in unanticipated drug-drug interactions that may cause or confound the assessment of toxicity. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the- counter medicine or herbal product. For information on CYP substrates and P-gp inhibitors or inducers see section 5.8.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form (including benzamide) of the investigational medicinal product
* Participation in other ongoing clinical trials.
* Pregnant or lactating females.
* Presence of underlying medical condition (e.g. gastrointestinal disorders or electrolyte disturbances) that in the opinion of the Investigator or Sponsor could adversely affect the ability of the subject to comply with or tolerate study procedures and/or study therapy, or confound the ability to interpret the tolerability of combined administration of entinostat and nivolumab in treated subjects
* Patients receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. The use of physiologic doses of corticosteroids (up to 5 mg/m2/day prednisone equivalent) may be approved after consultation with the Sponsor. No patient will be allowed to enroll in this trial more than once.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 91 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Dose Limiting Toxicity (DLT) of the combination treatment. | 5 weeks
  A dose limiting toxicity (DLT) is defined as any AE according to the definitions and exceptions listed below that is related to the administration of the combination of investigational agents occurring during the priming week and first cycle of combination treatment (first 5 weeks) in phase I of the trial.
  A study participant will be considered evaluable for a DLT if at least 2 doses of nivolumab and 4 doses of entinostat were administered during the first 5 weeks (5 weeks normally incorporate the priming week and 1 cycle of planned combination treatment). Participants who discontinue treatment or have treatment delays preventing them from receiving the above defined minimal amount of treatment in the first cycle of combination treatment for reasons unrelated to study drug toxicity, are not evaluable for DLT and will be replaced in enrollment (maximum number of replacement subjects will be 3 per dose level).
Phase II: Best response (CR or PR) | Change in 24 weeks
  Best response (CR or PR) will be based on RANO criteria for all primary CNS tumors and RECIST for non-CNS tumors, defined for each patient as the best response under study combination therapy during the first 6 cycles (assessment every 2 cycles).
  Calcified or intra-osseous (osteo)sarcoma target lesions which were progressive before initiation of treatment and show SD on response evaluation (confirmation through a subsequent scan at least 4 weeks later) will be considered as a responder.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Phase II: maximum of 48 weeks
  DOR will be evaluated for all patients who experienced (confirmed) response. Starting time point will be the time when best response was determined.
Disease Control Rate (DCR) | Phase II: maximum of 48 weeks
  DCR will be evaluated in addition, also using iRECIST and iRANO.
Stable disease (SD) | Phase II: maximum of 12 cycles (each cycle is 28 days)
  SD will be evaluated in addition, also using iRECIST and iRANO.
Progression-free survival (PFS) | 4 years
  The event-time endpoint PFS will be estimated using the Kaplan-Meier method, considering all the patients who started the treatment, whatever their compliance to treatment, including if the treatment was stopped prematurely for a reason other than disease progression. 95%-Confidence intervals will be provided for the Kaplan-Meier estimates.
Time to Response (TTR) | Phase II: maximum of 12 cycles (each cycle is 28 days)
  The event-time endpoint TTR will be estimated using the Kaplan-Meier method, considering all the patients who started the treatment, whatever their compliance to treatment, including if the treatment was stopped prematurely for a reason other than disease progression. 95%-Confidence intervals will be provided for the Kaplan-Meier estimates.
Overall Survival (OS) | Phase II: maximum of 48 weeks
  The event-time endpoint OS will be estimated using the Kaplan-Meier method, considering all the patients who started the treatment, whatever their compliance to treatment, including if the treatment was stopped prematurely for a reason other than disease progression. 95%-Confidence intervals will be provided for the Kaplan-Meier estimates.
Immune related Response Rate (RR) measured by iRECIST criteria and iRANO criteria | Phase II: maximum of 48 weeks
  As a secondary endpoint for patients who continued treatment beyond progression in case of clinical benefit, response as assessed by iRECIST or iRANO will be performed.
Maximum Plasma Time (Tmax) | one week
  Time to reach the maximum concentration (hr).
Maximum Plasma Concentration (Cmax) | one week
  The peak plasma concentration of a drug after Administration (ng/mL)
Half-life | one week
  The time required for the concentration of the drug to reach half of its original value (hr)
Area under the curve (AUC) | one week
  The integral of the concentration-time curve (ng/mL·hr)
total Clearance (CI/F) | one week
  The total body clearance will be equal to the renal clearance + hepatic clearance + lung clearance (L/h/m²)

OTHER OUTCOMES:
Exploratory: circulating tumor DNA (ctDNA) | At baseline and every odd cycle (Cycle 3 - 12) and every third cycle (Cycle 13 - 24) (each cycle is 28 days).
  Assessment of circulating Tumor DNA in peripheral blood.
Exploratory: Response prediction | 4 years
  Response prediction in a co-clinical PDX model and drug testing program
Exploratory: Immune phenotyping (FACS Panel) and Luminex cytokine panel | At baseline, after the priming week and after 5 weeks of initiation of therapy
  Immune phenotyping (FACS Panel) and Luminex cytokine panel in peripheral blood.
Exploratory: mRNA expression | 4 years
  Analyze mRNA Expression data for Tumor infiltrating immune cell populations
Exploratory: gene signatures | 4 years
  Analyze gene signature in whole exome data
Exploratory: cryptic transcription start sites | At baseline, after priming week and after 5 weeks of initiation of therapy
  Test induction of cryptic transcription start sites
Exploratory: Single nucleotide variant (SNV) load | 4 years
  Determination of SNV load by different methods (WES, Panel-Seq)

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Witt, Principal Investigator — University Hospital Heidelberg
Locations (14):
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- St. Anna Children's Hospital, Vienna, Austria
- Institut Curie, Paris, France
- Germany (5):
  - Augsburg University Hospital, Augsburg
  - Charité University Medicine Berlin, Berlin
  - Essen University Hospital, Essen
  - Hannover Medical School, Hanover
  - Hopp Children's Cancer Center Heidelberg (KiTZ), Heidelberg
- Prinses Máxima Centrum, Utrecht, Netherlands
- Karolinska Institute, Stockholm, Sweden
- Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The pseudonymized data will be shared for transparency reasons in the context of publications and after publication with other physicians and scientists (national and international academia) to promote and accelerate research on causes and treatment development of oncological diseases.
  Requests for access to pseudonymized patient data for non-INFORM-related scientific purposes will be reviewed by a Data Access Committee consisting of the INFORM Board, and the participating investigators. A positive statement of the respective ethic committee and a signed data protection commitment are requested. Requests should be addressed to the coordinating investigator Prof. Olaf Witt. Results of scientific research based on the INFORM2 NivEnt data may be used for academic teaching, research and scientific publications or presentations at scientific meetings.
Supporting Information: CSR
Time Frame: CSR will be available latest 1 year after the study is concluded.
Access Criteria: The CSR will be available via CTIS.

REFERENCES:
- [Derived] van Tilburg CM, Witt R, Heiss M, Pajtler KW, Plass C, Poschke I, Platten M, Harting I, Sedlaczek O, Freitag A, Meyrath D, Taylor L, Balasubramanian GP, Jager N, Pfaff E, Jones BC, Milde T, Pfister SM, Jones DTW, Kopp-Schneider A, Witt O. INFORM2 NivEnt: The first trial of the INFORM2 biomarker driven phase I/II trial series: the combination of nivolumab and entinostat in children and adolescents with refractory high-risk malignancies. BMC Cancer. 2020 Jun 5;20(1):523. doi: 10.1186/s12885-020-07008-8. PMID 32503469